CLINICAL TRIAL: NCT05322018
Title: Validation of a Novel Digital Pain Measure, Faces Thermometer Scale (FTS) in a Swedish Dental Context
Brief Title: Validation of Faces Thermometer Scale (FTS)
Status: Recruiting | Type: Observational
Sponsor: Malmö University (Other)
Collaborators: Lund University (Other)
Responsible Party: Principal Investigator, Rikard Roxner, Principal Investigator, Malmö University
Other Study IDs: FO 2021/570
Record Dates: First submitted 2022-02-09; First posted 2022-04-11 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Faces Thermometer Scale (FTS) — The Faces Thermometer Scale (FTS) is a one-item measure with 11 numeric rating scale steps (0, no pain to 10, much pain). Each step is associated with different faces and colors. The app presents all information in text, sound, and picture. FTS is part of PicPecc, an application for mobile devices. The child/adolescent assesses their pain on a tablet by moving the finger on the scale and points to the color and face that represent their appraised level of pain.

SUMMARY:
The aim of this study is to evaluate validity and reliability of a novel digital pain measure tool, the Faces Thermometer Scale (FTS). Pain is commonly reported by children and adolescents undergoing dental treatment. Pain is also a strongly contributing factor in the development of Dental Fear and Anxiety (DFA). Professionals often underestimate the pain perceived by their patients. Self-report tools are seldom used to measure pain in a clinical setting, denying child patients the possibility to communicate their pain experiences.

The aim of this study is to evaluate validity and reliability of a digital self-report pain measure tool, the Faces Thermometer Scale (FTS). Children and adolescents (N=150) aged 8 to 17 years visiting a dental clinic will be asked to score their pain using three different self-report pain tools; FTS, Faces Pain Scale-Revised (FPS-R) and Color Analog Scale (CAS). The validity and reliability of FPS-R and CAS is long established and will therefore be used to evaluate the psychometric properties of FTS.

DETAILED DESCRIPTION:
BACKGROUND Pain is a personal experience influenced by biological, psychological, and social factors. Pain is more than the sum of activity in sensory neurons and therefore different from nociception (Raja et al., 2020). Pain due to dental treatments and procedures is commonly reported by children and adolescents (Ghanei et al., 2018). Dental treatments giving rise to pain is considered a strongly contributing factor in the development of Dental Fear and Anxiety (DFA) and Dental Behavioral Management Problems (DBMP) in children (Klingberg et al., 1994; Radaal et al., 2002). Several studies have pointed to professionals underestimating pain compared to the perceived pain as reported by children themselves (Beyer et al., 1990; Versloot et al., 2004). Self-report tools are seldom used to measure pain in the clinical setting, denying child patients the possibility to communicate their pain experiences. One study showed that validated pain measure tools were used in only 19 % of cases in post-anesthesia care (Hetland Smeland et al., 2018). These findings point to the importance of letting children report their own pain experiences using validated tools easily accessible and which also children are willing to use.

As every-day life becomes progressively more digital through the use of internet and mobile devices the need for a valid and reliable digital self-report pain measure has become apparent. The use of a digital tool would also provide possibilities for real-time pain measure and empower children and adolescents in making their pain heard and understood facilitating pain-management in the inpatient care as well as outside the clinical setting. Analog scales and tools previously used for measuring pain are not directly transferable to a digital format. Digital tools are also preferred by children themselves over paper versions of the same scale. (Wood et al., 2011) The Faces Thermometer Scale (FTS) is a newly devised digital self-report tool to assess the intensity of children's and adolescents' pain. The FTS uses a 0 to 10 metric, 0 representing no pain and 10 indicating much pain. Each individual metric on the numeric scale is associated with a face and a color. FTS is part of and available through the mobile application Pictorial Support in Person-Centred Care for Children (PicPecc), which can be downloaded from App Store or Google Play.

Faces Pain Scale-Revised (FPS-R) (Hicks et al., 2001) and Color Analog Scale (CAS) (McGrath et al., 1996) are two frequently used and established analog self-report tools used in different settings to measure pain in children and adolescents. FPS-R and CAS have previously demonstrated convergent and discriminative validity, except for children under 7 years of age (Tsze et al., 2013). The same study showed good responsivity and reliability for both tools. FPS-R and CAS will be used to evaluate the psychometric properties of FTS.

The aim of this study is to evaluate the validity and reliability of the newly developed digital FTS tool for measuring children's pain. The hypotheses for this study are:

The FTS demonstrate an acceptable convergent validity in measuring pain in children aged 8-17, in relation to FPS-R and CAS.

The FTS shows acceptable constructive validity in measuring pain in children aged 8-17 in relation to FPS-R and CAS.

The FTS is reliable to use for pain measurement in children aged 8-17.

METHOD A consecutive sample of children and adolescents between the ages of 8 and 17 and meet the overall inclusion criteria are invited to participate in the study. The sample is drawn from patients visiting the pediatric general dental practice at the Faculty of Odontology at Malmö University. After inclusion, participants (N=150) are divided into four groups (no pain, acute pain, procedural pain, or postoperative pain/pain after surgery) depending on the presence of pain at inclusion and what type of procedure participants are scheduled for. Depending on these factors participants are asked about pain experience at between two to six times during the visit, using all three scales each time in a randomized order. Before first-time use, participants are introduced to each of the tools and familiarized on the use of each scale. FPS-R and CAS measurements are manually registered while pain measures on FTS are digitally recorded and stored.

We will determine the psychometric properties of FTS by analyzing convergent and construct validity/responsivity in relation to FPS-R and CAS. Comparative statistics will be employed but the exact statistical method to be used will be determined at a later stage and in cooperation with a statistician. Reliability will also be determined, even if not a measure of validity but a condition for a tool to be valid.

KNOWLEDGE GAINS The need for an easily available and valid mean for children to give voice to their pain experiences has become apparent. Evaluating the psychometric properties of the Faces Thermometer Scale (FTS) and thus validating a novel digital scale for measuring pain in children and adolescents will provide dental practitioners and researchers with such a tool.

ELIGIBILITY:
Inclusion Criteria:

* 8 to 17 years of age, undergoing dental procedures and/or examinations

Exclusion Criteria:

* cannot understand Swedish nor instructions on how to use the pain measure tools

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children and adolescents, 8 to 17 years of age, undergoing dental procedures and/or examinations
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Faces Thermometer Scale | Change in pain at up to 4 hours
  The Faces Thermometer Scale is a digital pain measure tool, which allows individuals to rate pain on a scale from 0 to 10 at intervals of 1. A higher reading indicates higher pain intensity.

SECONDARY OUTCOMES:
Faces Pain Scale-Revised | Change in pain at up to 4 hours
  The Faces Pain Scale-Revised is an analog pain measure tool, which allows individuals to rate pain on a scale from 0 to 10 at intervals of 2. A higher reading indicates higher pain intensity.
Color Analog Scale | Change in pain at up to 4 hours
  The Color Analog Scale is an analog pain measure tool, which allows individuals to rate pain on a continuous scale, which for the observer corresponds to a scale from 0 to 10 at intervals of 0.25. A higher reading indicates higher pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Gunilla Klingberg, Professor, Study Chair — Malmö University
Locations (1):
- Malmö University, Malmo, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ghanei M, Arnrup K, Robertson A. Procedural pain in routine dental care for children: a part of the Swedish BITA study. Eur Arch Paediatr Dent. 2018 Oct;19(5):365-372. doi: 10.1007/s40368-018-0368-2. Epub 2018 Sep 7. PMID 30194611
- [Background] Smeland AH, Twycross A, Lundeberg S, Rustoen T. Nurses' Knowledge, Attitudes and Clinical Practice in Pediatric Postoperative Pain Management. Pain Manag Nurs. 2018 Dec;19(6):585-598. doi: 10.1016/j.pmn.2018.04.006. Epub 2018 May 16. PMID 29778756
- [Background] Hicks CL, von Baeyer CL, Spafford PA, van Korlaar I, Goodenough B. The Faces Pain Scale-Revised: toward a common metric in pediatric pain measurement. Pain. 2001 Aug;93(2):173-183. doi: 10.1016/S0304-3959(01)00314-1. PMID 11427329
- [Background] Klingberg G, Vannas Lofqvist L, Bjarnason S, Noren JG. Dental behavior management problems in Swedish children. Community Dent Oral Epidemiol. 1994 Jun;22(3):201-5. doi: 10.1111/j.1600-0528.1994.tb01841.x. PMID 8070250
- [Background] McGrath PA, Seifert CE, Speechley KN, Booth JC, Stitt L, Gibson MC. A new analogue scale for assessing children's pain: an initial validation study. Pain. 1996 Mar;64(3):435-443. doi: 10.1016/0304-3959(95)00171-9. PMID 8783307
- [Background] Raadal M, Strand GV, Amarante EC, Kvale G. Relationship between caries prevalence at 5 years of age and dental anxiety at 10. Eur J Paediatr Dent. 2002 Mar;3(1):22-6. PMID 12871013
- [Background] Raja SN, Carr DB, Cohen M, Finnerup NB, Flor H, Gibson S, Keefe FJ, Mogil JS, Ringkamp M, Sluka KA, Song XJ, Stevens B, Sullivan MD, Tutelman PR, Ushida T, Vader K. The revised International Association for the Study of Pain definition of pain: concepts, challenges, and compromises. Pain. 2020 Sep 1;161(9):1976-1982. doi: 10.1097/j.pain.0000000000001939. PMID 32694387
- [Background] Tsze DS, von Baeyer CL, Bulloch B, Dayan PS. Validation of self-report pain scales in children. Pediatrics. 2013 Oct;132(4):e971-9. doi: 10.1542/peds.2013-1509. Epub 2013 Sep 2. PMID 23999954
- [Background] Versloot J, Veerkamp JS, Hoogstraten J. Assessment of pain by the child, dentist, and independent observers. Pediatr Dent. 2004 Sep-Oct;26(5):445-9. PMID 15460301
- [Background] Wood C, von Baeyer CL, Falinower S, Moyse D, Annequin D, Legout V. Electronic and paper versions of a faces pain intensity scale: concordance and preference in hospitalized children. BMC Pediatr. 2011 Oct 12;11:87. doi: 10.1186/1471-2431-11-87. PMID 21989306
- [Background] Beyer JE, McGrath PJ, Berde CB. Discordance between self-report and behavioral pain measures in children aged 3-7 years after surgery. J Pain Symptom Manage. 1990 Dec;5(6):350-6. doi: 10.1016/0885-3924(90)90029-j. PMID 2269802